CLINICAL TRIAL: NCT02513589
Title: Molecular Imaging of Inflammation With 18F-PBR06 to Identify Unstable Carotid Plaques in Patients With Stroke
Acronym: PLAQINSTEP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Negativity of the first results of in vivo binding of 18F-PBR06
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2014/17
Record Dates: First submitted 2015-07-30; First posted 2015-07-31 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Stroke
Keywords: Positron emission tomography; Carotid plaque; Inflammation; Stroke
MeSH Terms: conditions — Stroke; Inflammation | interventions — N-fluoroacetyl-N-(2,5-dimethoxybenzyl)-2-phenoxyaniline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Drug: 18F-PBR06

INTERVENTIONS:
Drug: 18F-PBR06 — Positron Emission Tomography / Computed Tomography (PET-CT) using 18F-PBR06

SUMMARY:
Evaluating an innovative molecular imaging technique to visualize inflammation of the atherosclerotic plaque in patients with a recent ischemic stroke (<15 days) with carotid stenosis> 50%, by performing a Positron emission tomography-computed tomography (PET-CT) with PBR06 18F, a tracer for Translocator protein (TPSO).

DETAILED DESCRIPTION:
More than one third of cerebral ischemic events are related to an atheromatous plaque. Inflammation, through a key player, the macrophage, is associated with increased metabolic activity of atherosclerotic plaque and its possible rupture. Inflammation within the plate is thus a marker of instability. These data underscore the importance of a prospective evaluation of inflammation with specific imaging with PET tracers inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Man with transient ischemic attack or recent ischemic stroke (<15j) in the carotid territory, confirmed by MRI
* Man with carotid stenosis> 50% on the side of stroke
* Male candidate for carotid endarterectomy
* Subject affiliated or beneficiary of a social security scheme
* Informed written consent

Exclusion Criteria:

* Women
* Chronic inflammatory disease in progress (cancer, vasculitis, ...)
* Patient with infection within 7 days
* A person placed under judicial protection, guardianship
* Incapable of giving consent
* Low affinity binder for TSPO

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Correlation between the value of standardized uptake value (SUV) on PET-CT with 18F-PBR06 and the degree of macrophage infiltration at histological examination | 15 days

SECONDARY OUTCOMES:
Levels of leukocyte and T lymphocyte inflammation of the plaque | 15 days
  Evaluate the constitutive parameters of the plaque (surface area, thickness, necrotic core and fibrous cap)
Plaque parameters composite | 15 days
  Evaluate the constitutive parameters of the plaque (surface area, thickness, necrotic core and fibrous cap)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo ZANOTTI-FREGONARA, Principal Investigator — University Hospital, Bordeaux; Paul Perez, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Schollhammer R, Lepreux S, Barthe N, Vimont D, Rullier A, Sibon I, Berard X, Zhang A, Kimura Y, Fujita M, Innis RB, Zanotti-Fregonara P, Morgat C. In vitro and pilot in vivo imaging of 18 kDa translocator protein (TSPO) in inflammatory vascular disease. EJNMMI Res. 2021 May 5;11(1):45. doi: 10.1186/s13550-021-00786-7. PMID 33950298